CLINICAL TRIAL: NCT04019964
Title: Nivolumab as a Non-Castrating Therapy for MMR-deficient and CDK12- Altered Prostate Cancer With PSA Recurrence After Local Therapy
Brief Title: Nivolumab in Biochemically Recurrent dMMR Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1933; IRB00205266 (Other: JHM IRB); CA209-76M (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2019-07-11; First posted 2019-07-15 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Prostate Cancer; Recurrent Prostate Cancer
Keywords: Prostate cancer; MMR-deficient prostate cancer; Biochemically recurrent prostate cancer; non-castrating therapy; Nivolumab
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab in biochemically recurrent prostate cancer (Experimental): Participants with previous prostatectomy or radiation therapy who subsequently developed detectable prostate specific antigen (PSA) levels ("biochemically recurrent prostate cancer").
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab 480mg intravenously every 4 weeks
  Other Names: Opdivo

SUMMARY:
MMR-deficient cancers of any histologic type appear to be very sensitive to PD-1 blockade with pembrolizumab, and similar data are also beginning to emerge for nivolumab and other immune checkpoint inhibitors. Among the MMR-deficient cancers, the best antitumor responses are often associated with high microsatellite instability (MSI-H status), higher tumor mutational burden (TMB), and higher predicted neoantigen load. Prevalence estimates of MMR deficiency across solid tumor types range from 1% to 20% depending on the type of malignancy. In prostate cancer, 1-3% of unselected cases harbor MMR deficiency and/or microsatellite instability.

For men who previously received definitive treatment for prostate cancer and subsequently develop detectable prostate specific antigen (PSA) levels, the clinical state is known as biochemically recurrent prostate cancer. The current standard of care treatment for patients with biochemically recurrent prostate cancer is either surveillance or androgen deprivation therapy (ADT). ADT has not been shown to provide a survival benefit in this setting, and the decision to initiate ADT will depend on patient preference and perceived risks of the disease. A non-hormonal therapy such as nivolumab would provide an alternative to ADT in patients with biomarker selected (i.e. dMMR, MSI-H, high TMB, or CDK12-altered) biochemically recurrent prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide signed informed consent and HIPAA authorization for the release of personal health information
* Males aged 18 years and above
* Prior local therapy with prostatectomy or EBRT/brachytherapy is required
* Prior salvage or adjuvant radiation therapy is allowed but not mandated. Radiation therapy must have been completed for at least 6 months.
* Absolute PSA >=1.0 ng/mL at screening
* Must have at least one of the following genetic alterations identified using archival tissue (i.e. prostate needle biopsy prior to radiation therapy or prostatectomy specimen):

  * Microsatellite instability (MSI-high) status by clinical grade testing
  * MMR protein loss (MSH2, MSH6, MLH1, PMS2) by immunohistochemistry
  * Inactivating mutation of MSH2, MSH6, MLH1 or PSM2 by clinical grade genomic testing
  * Tumor mutational burden >= 20 mutations/megabase (TMB >=20 muts/Mb) by clinical grade testing
  * Inactivating mutation (at least monoallelic of CDK12 by clinical grade testing
* Serum testosterone >= 150 ng/dL
* No radiographic evidence of metastatic disease by CT scan and bone scan, performed within the prior 4 weeks.
* Karnofsky Performance Status (KPS) >= 70% within 14 days before start of study treatment (ECOG <=1)
* Participants must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment as defined below:

  * Hemoglobin >= 9.0 g/dL with no blood transfusion in the past 28 days
  * Absolute neutrophil count (ANC) >= 1.0x10^9 / L
  * Platelet count >= 100 x 10^9 /L
  * Total bilirubin within institutional upper limit of normal (ULN) (in patients with Gilbert's syndrome, total bilirubin <1.5x institutional ULN will be acceptable)
  * Aspartate aminotransferase (AST), Serum Glutamic Oxaloacetic Transaminase (SGOT) / Alanine aminotransferase (ALT), Serum Glutamic Pyruvate Transaminase (SGPT) within institutional ULN
  * Participants must have creatinine clearance estimated using the Cockcroft-Gault equation of >=40 mL/min:

Estimated creatinine clearance = [(140 - age (years)) x weight (kg)] / [serum creatinine (mg/dL) x 72]

* Participants must have a life expectancy of >= 6 months
* Male participants and their partners who are sexually active and of childbearing potential must agree to the use of two highly effective forms of contraception in combination, throughout the period of taking study treatment and for 7 months after the last dose of nivolumab to prevent pregnancy in a partner.
* No evidence (within 5 years) of prior malignancies (except successfully treated basal cell or squamous cell carcinoma of the skin)

Exclusion Criteria:

* Metastatic disease or currently active second malignancy
* Prior androgen deprivation therapy (ADT) in the past 6 months. Prior ADT in context of neoadjuvant/adjuvant primary; prior ADT for biochemical recurrence is allowed, as long as no ADT has been administered in past 6 months and testosterone has recovered (>150 ng/dL)
* Prior oral anti-androgen (e.g. bicalutamide, nilutamide, enzalutamide, apalutamide), or androgen synthesis inhibitor (e.g. abiraterone, orteronel) within the past 2 weeks is not permitted. 5-alpha reductase inhibitor therapy (e.g. finasteride, dutasteride) is allowed, as long as subject has been stable on medication for past 6 months.
* Involvement in the planning and/or conduct of the study (applies to both BMS staff and/or staff at the study site)
* Participation in another clinical study with an investigational product during the last 4 weeks/28 days
* Patients should be excluded if they have had prior systemic treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways
* Patients should be excluded if they have an active, known or suspected autoimmune disease (e.g. inflammatory bowel disease, rheumatoid arthritis, autoimmune hepatitis, lupus, celiac disease). Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recure in the absence of an external trigger.
* Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone daily equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses >10mg daily prednisone equivalents are permitted in the absence of active autoimmune disease
* Permitted therapies include topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). Physiologic replacement doses of systemic corticosteroids are permitted, even if > 10 mg/day prednisone equivalents. A brief course of corticosteroids for prophylaxis (e.g. contrast dye allergy) or for treatment of nonautoimmune conditions (e.g. delayed-type hypersensitivity reaction caused by contact allergen) is permitted.
* As there is potential for hepatic toxicity with nivolumab, drugs with a predisposition to hepatotoxicity should be used with caution in patients treated with nivolumab-containing regimen.
* Patients should be excluded if they have a positive test for hepatitis B virus surface antigen (HBVsAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection
* Patients should be excluded if they have known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
* History of allergy to study drug components
* History of severe hypersensitivity reaction to any monoclonal antibody
* Any other serious illness or medical condition that would, in the opinion of the investigator, make this protocol unreasonably hazardous, including but not limited to:

  * Any uncontrolled major infection
  * Cardiac failure NYHA (New York Heart Association) III or IV
  * Crohn's disease or ulcerative colitis
  * Bone marrow dysplasia
  * Known allergy to any of the compounds under investigation
  * Unmanageable fecal incontinence
* Poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 6 months) myocardial infarction, uncontrolled major seizure disorder, extensive interstitial bilateral lung disease, or any psychiatric disorder that prohibits obtaining informed consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2025-04-23 (Actual); Study Completion 2025-07-03 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with PSA50 response | up to 6 months post-intervention
  Percentage of participants who have received at least 1 dose of Nivolumab who experience a confirmed >=50% decline in prostate specific antigen (PSA) from baseline, as defined by Prostate Cancer Working Group 3 (PCWG3) criteria.

SECONDARY OUTCOMES:
PSA progression-free survival (PSA-PFS) | up to 6 months post-intervention
  Median time from initiation of therapy until confirmed PSA increase of 25% (PCWG3). Estimated using Kaplan-Meier method.
Number of participants who achieve undetectable PSA | up to 6 months post-intervention
  Number of participants who achieve PSA < 0.1 ng/mL lasting at least 12 weeks.
Metastasis-free survival | up to 6 months post-intervention
  Median time from first dose of nivolumab until the development of radiographic metastatic disease on CT imaging and/or bone scan, as defined by PCWG3
Time to initiation of next systemic therapy | up to 6 months post-intervention
  Median time from first dose of nivolumab until next systemic therapy
Safety and tolerability of Nivolumab in biochemically recurrent prostate cancer as assessed by Incidence of Treatment-Emergent Adverse Events | up to 100 days post-intervention
  Number of participants experiencing adverse events Grade 3 or higher as defined by CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Mark Markowski, MD/PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2016. CA Cancer J Clin. 2016 Jan-Feb;66(1):7-30. doi: 10.3322/caac.21332. Epub 2016 Jan 7. PMID 26742998
- [Background] Scher HI, Morris MJ, Stadler WM, Higano C, Basch E, Fizazi K, Antonarakis ES, Beer TM, Carducci MA, Chi KN, Corn PG, de Bono JS, Dreicer R, George DJ, Heath EI, Hussain M, Kelly WK, Liu G, Logothetis C, Nanus D, Stein MN, Rathkopf DE, Slovin SF, Ryan CJ, Sartor O, Small EJ, Smith MR, Sternberg CN, Taplin ME, Wilding G, Nelson PS, Schwartz LH, Halabi S, Kantoff PW, Armstrong AJ; Prostate Cancer Clinical Trials Working Group 3. Trial Design and Objectives for Castration-Resistant Prostate Cancer: Updated Recommendations From the Prostate Cancer Clinical Trials Working Group 3. J Clin Oncol. 2016 Apr 20;34(12):1402-18. doi: 10.1200/JCO.2015.64.2702. Epub 2016 Feb 22. PMID 26903579
- [Background] Bubley GJ, Carducci M, Dahut W, Dawson N, Daliani D, Eisenberger M, Figg WD, Freidlin B, Halabi S, Hudes G, Hussain M, Kaplan R, Myers C, Oh W, Petrylak DP, Reed E, Roth B, Sartor O, Scher H, Simons J, Sinibaldi V, Small EJ, Smith MR, Trump DL, Wilding G, et al. Eligibility and response guidelines for phase II clinical trials in androgen-independent prostate cancer: recommendations from the Prostate-Specific Antigen Working Group. J Clin Oncol. 1999 Nov;17(11):3461-7. doi: 10.1200/JCO.1999.17.11.3461. PMID 10550143
- [Background] Stephenson AJ, Scardino PT, Kattan MW, Pisansky TM, Slawin KM, Klein EA, Anscher MS, Michalski JM, Sandler HM, Lin DW, Forman JD, Zelefsky MJ, Kestin LL, Roehrborn CG, Catton CN, DeWeese TL, Liauw SL, Valicenti RK, Kuban DA, Pollack A. Predicting the outcome of salvage radiation therapy for recurrent prostate cancer after radical prostatectomy. J Clin Oncol. 2007 May 20;25(15):2035-41. doi: 10.1200/JCO.2006.08.9607. PMID 17513807
- [Background] Nguyen T, Boldt RG, Rodrigues G. Prognostic Factors for Prostate Cancer Endpoints Following Biochemical Failure: A Review of the Literature. Cureus. 2015 Jan 5;7(1):e238. doi: 10.7759/cureus.238. eCollection 2015 Jan. PMID 26180662
- [Background] Antonarakis ES, Feng Z, Trock BJ, Humphreys EB, Carducci MA, Partin AW, Walsh PC, Eisenberger MA. The natural history of metastatic progression in men with prostate-specific antigen recurrence after radical prostatectomy: long-term follow-up. BJU Int. 2012 Jan;109(1):32-9. doi: 10.1111/j.1464-410X.2011.10422.x. Epub 2011 Jul 20. PMID 21777360
- [Background] Dong H, Strome SE, Salomao DR, Tamura H, Hirano F, Flies DB, Roche PC, Lu J, Zhu G, Tamada K, Lennon VA, Celis E, Chen L. Tumor-associated B7-H1 promotes T-cell apoptosis: a potential mechanism of immune evasion. Nat Med. 2002 Aug;8(8):793-800. doi: 10.1038/nm730. Epub 2002 Jun 24. PMID 12091876
- [Background] Wintterle S, Schreiner B, Mitsdoerffer M, Schneider D, Chen L, Meyermann R, Weller M, Wiendl H. Expression of the B7-related molecule B7-H1 by glioma cells: a potential mechanism of immune paralysis. Cancer Res. 2003 Nov 1;63(21):7462-7. PMID 14612546
- [Background] Dong H, Chen L. B7-H1 pathway and its role in the evasion of tumor immunity. J Mol Med (Berl). 2003 May;81(5):281-7. doi: 10.1007/s00109-003-0430-2. Epub 2003 Apr 30. PMID 12721664
- [Background] Pardoll DM. The blockade of immune checkpoints in cancer immunotherapy. Nat Rev Cancer. 2012 Mar 22;12(4):252-64. doi: 10.1038/nrc3239. PMID 22437870
- [Background] Thompson RH, Gillett MD, Cheville JC, Lohse CM, Dong H, Webster WS, Krejci KG, Lobo JR, Sengupta S, Chen L, Zincke H, Blute ML, Strome SE, Leibovich BC, Kwon ED. Costimulatory B7-H1 in renal cell carcinoma patients: Indicator of tumor aggressiveness and potential therapeutic target. Proc Natl Acad Sci U S A. 2004 Dec 7;101(49):17174-9. doi: 10.1073/pnas.0406351101. Epub 2004 Nov 29. PMID 15569934
- [Background] Thompson RH, Gillett MD, Cheville JC, Lohse CM, Dong H, Webster WS, Chen L, Zincke H, Blute ML, Leibovich BC, Kwon ED. Costimulatory molecule B7-H1 in primary and metastatic clear cell renal cell carcinoma. Cancer. 2005 Nov 15;104(10):2084-91. doi: 10.1002/cncr.21470. PMID 16208700
- [Background] Thompson RH, Kuntz SM, Leibovich BC, Dong H, Lohse CM, Webster WS, Sengupta S, Frank I, Parker AS, Zincke H, Blute ML, Sebo TJ, Cheville JC, Kwon ED. Tumor B7-H1 is associated with poor prognosis in renal cell carcinoma patients with long-term follow-up. Cancer Res. 2006 Apr 1;66(7):3381-5. doi: 10.1158/0008-5472.CAN-05-4303. PMID 16585157
- [Background] Ohigashi Y, Sho M, Yamada Y, Tsurui Y, Hamada K, Ikeda N, Mizuno T, Yoriki R, Kashizuka H, Yane K, Tsushima F, Otsuki N, Yagita H, Azuma M, Nakajima Y. Clinical significance of programmed death-1 ligand-1 and programmed death-1 ligand-2 expression in human esophageal cancer. Clin Cancer Res. 2005 Apr 15;11(8):2947-53. doi: 10.1158/1078-0432.CCR-04-1469. PMID 15837746
- [Background] Wu C, Zhu Y, Jiang J, Zhao J, Zhang XG, Xu N. Immunohistochemical localization of programmed death-1 ligand-1 (PD-L1) in gastric carcinoma and its clinical significance. Acta Histochem. 2006;108(1):19-24. doi: 10.1016/j.acthis.2006.01.003. Epub 2006 Mar 13. PMID 16530813
- [Background] Nomi T, Sho M, Akahori T, Hamada K, Kubo A, Kanehiro H, Nakamura S, Enomoto K, Yagita H, Azuma M, Nakajima Y. Clinical significance and therapeutic potential of the programmed death-1 ligand/programmed death-1 pathway in human pancreatic cancer. Clin Cancer Res. 2007 Apr 1;13(7):2151-7. doi: 10.1158/1078-0432.CCR-06-2746. PMID 17404099
- [Background] Zitvogel L, Tesniere A, Kroemer G. Cancer despite immunosurveillance: immunoselection and immunosubversion. Nat Rev Immunol. 2006 Oct;6(10):715-27. doi: 10.1038/nri1936. Epub 2006 Sep 15. PMID 16977338
- [Background] Taube JM, Anders RA, Young GD, Xu H, Sharma R, McMiller TL, Chen S, Klein AP, Pardoll DM, Topalian SL, Chen L. Colocalization of inflammatory response with B7-h1 expression in human melanocytic lesions supports an adaptive resistance mechanism of immune escape. Sci Transl Med. 2012 Mar 28;4(127):127ra37. doi: 10.1126/scitranslmed.3003689. PMID 22461641
- [Background] Iwai Y, Terawaki S, Honjo T. PD-1 blockade inhibits hematogenous spread of poorly immunogenic tumor cells by enhanced recruitment of effector T cells. Int Immunol. 2005 Feb;17(2):133-44. doi: 10.1093/intimm/dxh194. Epub 2004 Dec 20. PMID 15611321
- [Background] Hirano F, Kaneko K, Tamura H, Dong H, Wang S, Ichikawa M, Rietz C, Flies DB, Lau JS, Zhu G, Tamada K, Chen L. Blockade of B7-H1 and PD-1 by monoclonal antibodies potentiates cancer therapeutic immunity. Cancer Res. 2005 Feb 1;65(3):1089-96. PMID 15705911
- [Background] Li B, VanRoey M, Wang C, Chen TH, Korman A, Jooss K. Anti-programmed death-1 synergizes with granulocyte macrophage colony-stimulating factor--secreting tumor cell immunotherapy providing therapeutic benefit to mice with established tumors. Clin Cancer Res. 2009 Mar 1;15(5):1623-34. doi: 10.1158/1078-0432.CCR-08-1825. Epub 2009 Feb 10. PMID 19208793
- [Background] Curran MA, Montalvo W, Yagita H, Allison JP. PD-1 and CTLA-4 combination blockade expands infiltrating T cells and reduces regulatory T and myeloid cells within B16 melanoma tumors. Proc Natl Acad Sci U S A. 2010 Mar 2;107(9):4275-80. doi: 10.1073/pnas.0915174107. Epub 2010 Feb 16. PMID 20160101
- [Background] Beer TM, Kwon ED, Drake CG, Fizazi K, Logothetis C, Gravis G, Ganju V, Polikoff J, Saad F, Humanski P, Piulats JM, Gonzalez Mella P, Ng SS, Jaeger D, Parnis FX, Franke FA, Puente J, Carvajal R, Sengelov L, McHenry MB, Varma A, van den Eertwegh AJ, Gerritsen W. Randomized, Double-Blind, Phase III Trial of Ipilimumab Versus Placebo in Asymptomatic or Minimally Symptomatic Patients With Metastatic Chemotherapy-Naive Castration-Resistant Prostate Cancer. J Clin Oncol. 2017 Jan;35(1):40-47. doi: 10.1200/JCO.2016.69.1584. Epub 2016 Oct 31. PMID 28034081
- [Background] Kwon ED, Drake CG, Scher HI, Fizazi K, Bossi A, van den Eertwegh AJ, Krainer M, Houede N, Santos R, Mahammedi H, Ng S, Maio M, Franke FA, Sundar S, Agarwal N, Bergman AM, Ciuleanu TE, Korbenfeld E, Sengelov L, Hansen S, Logothetis C, Beer TM, McHenry MB, Gagnier P, Liu D, Gerritsen WR; CA184-043 Investigators. Ipilimumab versus placebo after radiotherapy in patients with metastatic castration-resistant prostate cancer that had progressed after docetaxel chemotherapy (CA184-043): a multicentre, randomised, double-blind, phase 3 trial. Lancet Oncol. 2014 Jun;15(7):700-12. doi: 10.1016/S1470-2045(14)70189-5. Epub 2014 May 13. PMID 24831977
- [Background] Graff JN, Alumkal JJ, Drake CG, Thomas GV, Redmond WL, Farhad M, Cetnar JP, Ey FS, Bergan RC, Slottke R, Beer TM. Early evidence of anti-PD-1 activity in enzalutamide-resistant prostate cancer. Oncotarget. 2016 Aug 16;7(33):52810-52817. doi: 10.18632/oncotarget.10547. PMID 27429197
- [Background] Le DT, Uram JN, Wang H, Bartlett BR, Kemberling H, Eyring AD, Skora AD, Luber BS, Azad NS, Laheru D, Biedrzycki B, Donehower RC, Zaheer A, Fisher GA, Crocenzi TS, Lee JJ, Duffy SM, Goldberg RM, de la Chapelle A, Koshiji M, Bhaijee F, Huebner T, Hruban RH, Wood LD, Cuka N, Pardoll DM, Papadopoulos N, Kinzler KW, Zhou S, Cornish TC, Taube JM, Anders RA, Eshleman JR, Vogelstein B, Diaz LA Jr. PD-1 Blockade in Tumors with Mismatch-Repair Deficiency. N Engl J Med. 2015 Jun 25;372(26):2509-20. doi: 10.1056/NEJMoa1500596. Epub 2015 May 30. PMID 26028255
- [Background] Cortes-Ciriano I, Lee S, Park WY, Kim TM, Park PJ. A molecular portrait of microsatellite instability across multiple cancers. Nat Commun. 2017 Jun 6;8:15180. doi: 10.1038/ncomms15180. PMID 28585546
- [Background] Robinson D, Van Allen EM, Wu YM, Schultz N, Lonigro RJ, Mosquera JM, Montgomery B, Taplin ME, Pritchard CC, Attard G, Beltran H, Abida W, Bradley RK, Vinson J, Cao X, Vats P, Kunju LP, Hussain M, Feng FY, Tomlins SA, Cooney KA, Smith DC, Brennan C, Siddiqui J, Mehra R, Chen Y, Rathkopf DE, Morris MJ, Solomon SB, Durack JC, Reuter VE, Gopalan A, Gao J, Loda M, Lis RT, Bowden M, Balk SP, Gaviola G, Sougnez C, Gupta M, Yu EY, Mostaghel EA, Cheng HH, Mulcahy H, True LD, Plymate SR, Dvinge H, Ferraldeschi R, Flohr P, Miranda S, Zafeiriou Z, Tunariu N, Mateo J, Perez-Lopez R, Demichelis F, Robinson BD, Schiffman M, Nanus DM, Tagawa ST, Sigaras A, Eng KW, Elemento O, Sboner A, Heath EI, Scher HI, Pienta KJ, Kantoff P, de Bono JS, Rubin MA, Nelson PS, Garraway LA, Sawyers CL, Chinnaiyan AM. Integrative clinical genomics of advanced prostate cancer. Cell. 2015 May 21;161(5):1215-1228. doi: 10.1016/j.cell.2015.05.001. PMID 26000489
- [Background] Wu YM, Cieslik M, Lonigro RJ, Vats P, Reimers MA, Cao X, Ning Y, Wang L, Kunju LP, de Sarkar N, Heath EI, Chou J, Feng FY, Nelson PS, de Bono JS, Zou W, Montgomery B, Alva A; PCF/SU2C International Prostate Cancer Dream Team; Robinson DR, Chinnaiyan AM. Inactivation of CDK12 Delineates a Distinct Immunogenic Class of Advanced Prostate Cancer. Cell. 2018 Jun 14;173(7):1770-1782.e14. doi: 10.1016/j.cell.2018.04.034. PMID 29906450
- [Background] Antonarakis ES. Cyclin-Dependent Kinase 12, Immunity, and Prostate Cancer. N Engl J Med. 2018 Sep 13;379(11):1087-1089. doi: 10.1056/NEJMcibr1808772. No abstract available. PMID 30207914
- [Background] Abida W, Cheng ML, Armenia J, Middha S, Autio KA, Vargas HA, Rathkopf D, Morris MJ, Danila DC, Slovin SF, Carbone E, Barnett ES, Hullings M, Hechtman JF, Zehir A, Shia J, Jonsson P, Stadler ZK, Srinivasan P, Laudone VP, Reuter V, Wolchok JD, Socci ND, Taylor BS, Berger MF, Kantoff PW, Sawyers CL, Schultz N, Solit DB, Gopalan A, Scher HI. Analysis of the Prevalence of Microsatellite Instability in Prostate Cancer and Response to Immune Checkpoint Blockade. JAMA Oncol. 2019 Apr 1;5(4):471-478. doi: 10.1001/jamaoncol.2018.5801. PMID 30589920
- [Background] Long GV, Tykodi SS, Schneider JG, Garbe C, Gravis G, Rashford M, Agrawal S, Grigoryeva E, Bello A, Roy A, Rollin L, Zhao X. Assessment of nivolumab exposure and clinical safety of 480 mg every 4 weeks flat-dosing schedule in patients with cancer. Ann Oncol. 2018 Nov 1;29(11):2208-2213. doi: 10.1093/annonc/mdy408. PMID 30215677
- [Background] Therasse P, Arbuck SG, Eisenhauer EA, Wanders J, Kaplan RS, Rubinstein L, Verweij J, Van Glabbeke M, van Oosterom AT, Christian MC, Gwyther SG. New guidelines to evaluate the response to treatment in solid tumors. European Organization for Research and Treatment of Cancer, National Cancer Institute of the United States, National Cancer Institute of Canada. J Natl Cancer Inst. 2000 Feb 2;92(3):205-16. doi: 10.1093/jnci/92.3.205. PMID 10655437